CLINICAL TRIAL: NCT03533543
Title: A Retrospective Cohort Study on the Burden of New-Onset Atrial Fibrillation Complicating Acute Myocardial Infarction at Shanghai Tenth People's Hospital
Brief Title: New-Onset Atrial Fibrillation Complicating Acute Myocardial Infarction in ShangHai
Acronym: NOAFCAMI-SH
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Other Study IDs: NOAFCAMI-SH
Record Dates: First submitted 2018-04-28; First posted 2018-05-23 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation; Myocardial Infarction
Keywords: Myocardial infarction; New-onset atrial fibrillation; Retrospective; Prognosis
MeSH Terms: conditions — Atrial Fibrillation; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New-onset atrial fibrillation: Patients with MI who are free from a medical history of atrial fibrillation (AF) will be recognized as NOAF if they develop an atrial fibrillation (lasting for at least 30 seconds which are recorded by CEM) incident during hospitalization.
  Interventions: Device: CEM
- Non new-onset atrial fibrillation: Patients with MI who are free from a medical history of AF will be recognized as Non-NOAF if they persist with sinus rhythm (based on CEM) during hospitalization.
  Interventions: Device: CEM

INTERVENTIONS:
Device: CEM — All patients with MI hospitalized in the CCU department of Shanghai Tenth People's Hospital will receive 24-hour cardiac monitoring until discharge.

SUMMARY:
To characterize and estimate the incidence rate of new-onset atrial fibrillation (NOAF) in patients with acute myocardial infarction (MI). To explore the prognostic influences of NOAF on MI patients' clinical outcomes. To further investigate the impact of NOAF associated characteristics on patients' clinical outcomes eithier during hospitalization or follow-up period.

DETAILED DESCRIPTION:
In the present study, investigators retrospectively reviewed the medical records of all acute MI patients who were admitted to the coronary artery unit (CCU) of Shanghai Tenth People's Hospital between February 2014 and March 2018.

All eligible patients' demographics, cardiovascular risk factors, comorbidities, laboratory tests, echocardiography data, angiography data, acute and dischage medications, and clinical outcomes will be collected. All patients admitt to our CCU department will receive CEM immediately after admission and continue until discharge. Heart thythm status and those characteristics assoicated with NOAF will be reviewed by several independent physicians and recorded in a centralized electronic database.

Several post-MI NOAF assoicated characteristics and definitions are displayed as follows:

1. Total CEM duration is defined as the period during which the monitor was started after admission and turned off before discharge.
2. AF maintained duration is defined as the period during which an AF episode presented and terminated.
3. Total AF duration is calculated by summing all AF episodes' maintained durations descripted above.
4. AF burden was calculated by dividing the total AF duration by the total CEM duration.
5. NOAF pattern included paroxysmal NOAF, persistent NOAF, transient NOAF, and persisting NOAF, definitions are demonstrated as follows:

1) Paroxysmal NOAF is defined as more than 1 episodes of AF occur during hospitalization irrespective of the discharge rhythm status or only 1 episode of AF is observed during hospitalization and maintain sinus rhythm at discharge.

2) Persistent NOAF is defined as only 1 episode of AF is observed during hospitalization and maintain AF at discharge.

3) Transient NOAF is recorded if AF episodes only occur during hospitalization with emergency department ECG, on-admission ECG and discharge ECG maintaining sinus rhythm, irrespective of the frequencies of AF.

4) Persisting NOAF is recorded if AF episodes occur during hospitalization with a discharge ECG still maintaining AF rhythm, irrespective of the frequencies of AF.

6. Frequencies of NOAF

7. Symptomatic and silent NOAF

1. Symptomatic AF is defined as AFresulting in clinical symptoms or the need for urgent cardioversion.
2. Silent AF is defined as any asymptomatic episodes of AF lasting for over 30 seconds at CEM.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for acute MI between February 2014 and March 2018 in the CCU department of Shanghai Tenth People's Hospital;
* Adult patients (>18 years old).

Exclusion Criteria:

* Patients with a medical history of pre-existing AF;
* Patietns with a medical histroy of Rheumatic valvular disease;
* Patietns with a medical histroy of sick sinus syndrome;
* Patients undergoing emergent coronary artery bypass surgery;
* Patients' medical records with serious deficiencies and critical information (e.g. demographic data, laboratory testings, etc.) cannot be retrieved;
* Patients who refused to receive electronic monitoring during hospitalization and the data of cardiac rhythm cannot be obtained;
* Premature discharge due to nonmedical reasons such as nonpayment, failure to comply with program rules, conflicting with treatment staff, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute MI without a medical history of AF.
Sampling Method: Non-Probability Sample
Enrollment: 2399 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac event (MACE) | From the time of admission to coronary care unit until occurrence of an outcome of interest, death, loss to follow up or April 10, 2019, maximum up to 5 years
  Cardiovascular death, recurrent myocardial infarction, rehospitalization for heart failure or stroke

SECONDARY OUTCOMES:
All-cause death | From the time of admission to coronary care unit until occurrence of an outcome of interest, death, loss to follow up or April 10, 2019, maximum up to 5 years
  Death from any cause
Cardiovascular death | From the time of admission to coronary care unit until occurrence of an outcome of interest, death, loss to follow up or April 10, 2019, maximum up to 5 years
  Death from cardiovascular causes
Recurrent myocardial infarction | From the time of admission to coronary care unit until occurrence of an outcome of interest, death, loss to follow up or April 10, 2019, maximum up to 5 years
  Rehospitalization for myocardial infarction
Rehospitalization for heart failure | From the time of admission to coronary care unit until occurrence of an outcome of interest, death, loss to follow up or April 10, 2019, maximum up to 5 years
  Rehospitalization for heart failure
Stroke | From the time of admission to coronary care unit until occurrence of an outcome of interest, death, loss to follow up or April 10, 2019, maximum up to 5 years
  Stroke is defined as the presence of a new focal neurologic deficit thought to be vascular in origin, with signs or symptoms lasting>24h.
In-hospital MACE | 30 days
  Cardiovascular death, nonfatal re-infarction, new congestive heart failure or ischemic stroke at 30 days
In-hospital sustained ventricular tachycardia/ventricular fibrillation | From the time of admission to coronary care unit until discharge
  Sustianed ventricular tachycardia is defined as ventricular arrhythemia lasting for over 30s where emergent cardioversion is required. Ventricular fibrillation is defined as the heart quivers instead of pumping due to disorganized electrical activity in the ventricles.
In-hospital cardiogenic shock | From the time of admission to coronary care unit until discharge
  Cardiogenic shock is defined as systolic blood pressure < 90 mmHg not responsive to fluid resuscitation where IV intropes are required.
Nonfatal re-infarction at 30 days | 30 days
  Re-infarction is defined as recurrent ischemic symptoms> 20 min with new ST elevation> 0.1mV in≥ 2 contiguous leads and was verified by an urgent angiography.
Ischemic stroke at 30 days | 30 days
  Ischemic stroke is defined as the presence of a new focal neurologic deficit thought to be ischemic in origin, with signs or symptoms lasting over 24 hours, which is validated based on a computerized tomography (CT) or magnetic resonance imaging (MRI) examination.
New congestive heart failure at 30 days | 30 days
  New congestive heart failure is defined as the first episode of cardiac decompensation requiring intravenous diuretics when patients suffer chest distress, polypnea or dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Yidong Wei, MD, PhD, Principal Investigator — Department of Cardiology, Shanghai Tenth People's Hospital
Locations (1):
- Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Luo J, Xu S, Li H, Gong M, Li Z, Liu B, Qin X, Shi B, Wei Y. Long-term impact of the burden of new-onset atrial fibrillation in patients with acute myocardial infarction: results from the NOAFCAMI-SH registry. Europace. 2021 Feb 5;23(2):196-204. doi: 10.1093/europace/euaa234. PMID 32929491
- [Result] Luo J, Xu S, Li H, Li Z, Liu B, Qin X, Gong M, Shi B, Wei Y. Long-term impact of new-onset atrial fibrillation complicating acute myocardial infarction on heart failure. ESC Heart Fail. 2020 Oct;7(5):2762-2772. doi: 10.1002/ehf2.12872. Epub 2020 Jun 23. PMID 32578394
- [Result] Luo J, Liu B, Li H, Xu S, Gong M, Li Z, Qin X, Shi B, Hao C, Zhang J, Wei Y. Prognostic Impact of the Symptom of New-Onset Atrial Fibrillation in Acute Myocardial Infarction: Insights From the NOAFCAMI-SH Registry. Front Cardiovasc Med. 2021 Sep 22;8:677695. doi: 10.3389/fcvm.2021.677695. eCollection 2021. PMID 34631808
- [Result] Hao C, Luo J, Liu B, Xu W, Li Z, Gong M, Qin X, Shi B, Wei Y. Prognostic Significance of New-Onset Atrial Fibrillation in Heart Failure with Preserved, Mid-Range, and Reduced Ejection Fraction Following Acute Myocardial Infarction: Data from the NOAFCAMI-SH Registry. Clin Interv Aging. 2022 Apr 13;17:479-493. doi: 10.2147/CIA.S358349. eCollection 2022. PMID 35444413
- [Result] Luo J, Xu S, Li H, Li Z, Gong M, Qin X, Zhang X, Hao C, Liu X, Zhang W, Xu W, Liu B, Wei Y. Prognostic impact of stress hyperglycemia ratio in acute myocardial infarction patients with and without diabetes mellitus. Nutr Metab Cardiovasc Dis. 2022 Oct;32(10):2356-2366. doi: 10.1016/j.numecd.2022.07.004. Epub 2022 Jul 16. PMID 35965248
- [Result] Luo J, Li Z, Qin X, Zhang X, Liu X, Zhang W, Xu W, Zhang Y, Fang Y, Liu B, Wei Y; NOAFCAMI-SH Registry Investigators. Prognostic implications of the 4S-AF scheme to characterize new-onset atrial fibrillation after myocardial infarction. Eur J Intern Med. 2023 Jul;113:38-44. doi: 10.1016/j.ejim.2023.04.003. Epub 2023 Apr 8. PMID 37037721
- [Result] Luo J, Li Z, Qin X, Zhang X, Liu X, Zhang W, Xu W, Liu B, Wei Y; NOAFCAMI-SH Registry Investigators. Association of stress hyperglycemia ratio with in-hospital new-onset atrial fibrillation and long-term outcomes in patients with acute myocardial infarction. Diabetes Metab Res Rev. 2024 Feb;40(2):e3726. doi: 10.1002/dmrr.3726. Epub 2023 Sep 15. PMID 37712510
- [Result] Luo J, Qin X, Zhang X, Zhang Y, Yuan F, Shi W, Liu B, Wei Y; NOAFCAMI-SH Registry Investigators. Prognostic implications of systemic immune-inflammation index in myocardial infarction patients with and without diabetes: insights from the NOAFCAMI-SH registry. Cardiovasc Diabetol. 2024 Jan 22;23(1):41. doi: 10.1186/s12933-024-02129-x. PMID 38254086
- [Result] Luo J, Qin X, Zhang X, Zhang Y, Fang Y, Shi W, Liu B, Wei Y; NOAFCAMI-SH Registry Investigators. Prognostic impact of new-onset atrial fibrillation in myocardial infarction with and without improved ejection fraction. ESC Heart Fail. 2024 Dec;11(6):3713-3722. doi: 10.1002/ehf2.14956. Epub 2024 Jul 10. PMID 38984376